CLINICAL TRIAL: NCT02828813
Title: Neural Mechanisms of Motor and Cognitive Networks
Status: Completed | Type: Observational
Sponsor: National Research Center for Rehabilitation Technical Aids (Other)
Responsible Party: Principal Investigator, Pengxu Wei, Director, National Research Center for Rehabilitation Technical Aids
Other Study IDs: NRRA201607
Record Dates: First submitted 2016-07-05; First posted 2016-07-12 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Normal Volunteers; Cognition Disorders; Motor Disorders
MeSH Terms: conditions — Cognition Disorders; Motor Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Normal: healthy subjects
- CogImpair: persons with cognitive impairments
- MotorDeficits: persons with motor deficits

SUMMARY:
This study investigates the neural mechanisms of motor and cognitive networks using cognitive assessment, reaction time measurement, high-density EEG and fMRI.

ELIGIBILITY:
Inclusion Criteria (for healthy people):

* right handed,
* no history of psychological/psychotic problems,
* no history of important diseases.

Exclusion Criteria (for healthy people):

* Being Pregnant or breast feeding
* having any non-MRI compatible conditions

Inclusion Criteria (for patients):

* right handed
* in a stable condition
* ability to follow complex commands

Exclusion Criteria (for patients):

* having any non-MRI compatible conditions
* inability to perform required tasks

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy Volunteers: Advertising recruitment Persons with cognitive impairments: from inpatients and outpatients Persons with motor deficits: from inpatients and outpatients
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2016-06; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
cognitive assessment scores | within one week

OTHER OUTCOMES:
reaction time measurement | within one week
EEG | within one week
fMRI | within one week

CONTACTS AND LOCATIONS:
Overall Officials: PX Wei, Dr., Principal Investigator — National Research Center for Rehabilitation Technical Aids
Locations (1):
- National Research Center for Rehabilitation Technical Aids, Beijing, China

IPD SHARING:
Plan to Share IPD: No
no plan to share data